CLINICAL TRIAL: NCT01542840
Title: Onset Time of Ultrasound-Guided Popliteal Sciatic Nerve Block: Comparing Circumferential Injection of Local Anesthetic to Injection That Separates the Nerve in Its Two Components
Brief Title: Onset Time of Nerve Block: A Comparison of Two Injection Locations in Patients Having Lower Leg/ Foot Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Kristie Osteen, Anesthesiologist, Ochsner Health System
Other Study IDs: 2011.200.C
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Strain of Muscle and/or Tendon of Lower Leg; Fracture of Lower Leg; Crushing Injury of Lower Leg; Fracture Malunion - Ankle and/or Foot; Disorder of Joint of Ankle and/or Foot; Complete Tear, Ankle and/or Foot Ligament; Pathological Fracture - Ankle and/or Foot; Loose Body in Joint of Ankle and/or Foot
Keywords: surgery; orthopedic surgery; foot surgery; leg surgery; ankle surgery; leg; foot; ankle; anesthesia; local anesthesia; regional anesthesia; Ochsner Clinic; Ochsner Hospital; New Orleans; Louisiana; Kristie Osteen, MD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare injecting local anesthetic (numbing medication) in different patterns around a major nerve in the leg. Patients who undergo surgery to the lower leg and/or foot are usually offered the option of a nerve block to help with pain control after surgery. A nerve block involves injecting local anesthetic (numbing medicine) by a nerve or nerves that provide sensation to the area where surgery will be performed. The local anesthetic (numbing medication) numbs up the area where the surgery is performed and helps decrease the amount of pain felt after surgery. The local anesthetic (numbing medication) can be injected in various patterns by a nerve, such as in one spot by a nerve or completely surrounding a nerve. The local anesthetic will be either injected around the sciatic nerve or will injected in a way that will split the sciatic nerve into the two component nerves that make it up, the tibial and sciatic, and surrounds each nerve.

The hypothesis is that subjects in the group that local anesthetic is injected in a pattern that separates the sciatic nerve into the two component nerves may have a faster onset time of regional anesthesia and block success than subjects in the group that have the local anesthetic injected at around the nerve.

DETAILED DESCRIPTION:
After the consent form is signed, subjects will be randomly assigned (like the flip of a coin) to either receive the local anesthestic (numbing medication) around the sciatic nerve or in a pattern that separates the sciatic nerve into the two component nerves that make it up, the tibial and sciatic, and surrounds each nerve.

Before the nerve block is performed, the movement and sensation in the subject's foot will be checked to make sure it is normal. They will be asked to move their foot up and down. Using a blunt safety needle, their foot will be gently touched in different places to see if they can feel sharp sensations.

The amount of relaxation medication before the block will be recorded. The local anesthetic (numbing medication) will be injected in the pattern subjects were randomly assigned. The time it takes from the moment they are asked to say their name and birthday until they cannot move or feel their foot will be recorded.

Five minutes from the time the injection is complete, subjects will be asked to move their foot up and down. Also, their foot will be gently touched in different places with a blunt safety needle to see if they can still feel sharp sensations. Subjects will be asked to do this every five minutes until they cannot feel any sensation in their foot or if thirty minutes pass.

A member of the study team will contact subjects by telephone in about a week to see if they have any pain, numbness, and/or weakness in their leg/foot.

ELIGIBILITY:
Inclusion Criteria:

* undergoing lower leg and/or foot surgery
* ASA Physical status I-III
* ability to give informed consent
* age 18 years old or older

Exclusion Criteria:

* true allergy to local anesthetics, not sensitivity, as determined by investigator
* bilateral lower extremity surgery
* patient refusal
* infection at the injection site
* peripheral neuropathy of lower extremity as documented by electromyography studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing lower leg and/or foot surgery at Ochsner Clinic Foundation's Main Campus.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kristie D Osteen, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States